CLINICAL TRIAL: NCT00369434
Title: A Double-Blind, Randomized, Placebo-Controlled, Efficacy and Safety Study of DVS SR for Treatment of Vasomotor Symptoms Associated With Menopause
Brief Title: Study of the Safety and Efficacy of Desvenlafaxine Succinate for Vasomotor Symptoms in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A2-337
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Menopause; Vasomotor System

INTERVENTIONS:
Drug: Desvenlafaxine succinate sustained-release (DVS SR)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of 100 mg and 150 mg of DVS SR, an extended release form of desvenlafaxine succinate, in comparison to placebo for the treatment of Vasomotor Symptoms (VMS) associated with menopause in a population of postmenopausal women.

DETAILED DESCRIPTION:
To assess the efficacy and safety of 100 mg and 150 mg of DVS SR in comparison to placebo for the treatment of moderate to severe VMS associated with menopause, as well as additional outcome indicators such as sleep disruptions, overall climacteric symptoms, mood changes, somatic symptoms, and overall satisfaction with DVS SR in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women who seek treatment for hot flushes
* Body Mass Index (BMI) less than or equal to 40 kg/m2

Other inclusions apply.

Exclusion Criteria:

* Hypersensitivity to Venlafaxine
* Myocardial infarction and/or unstable angina within 6 months of screening
* History of seizure disorder

Other exclusions apply.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2006-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The number and severity of hot flushes collected throughout the study after 12 weeks of therapy.

SECONDARY OUTCOMES:
The number of awakenings due to VMS and the total mood disturbance score (Profile of Mood States [POMS]).
The scores on the Greene Climacteric Scale (GCS), the Visual Analog Scale-Pain Intensity (VAS-PI), and the Satisfaction Survey (SS).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (34):
- United States (34):
  - Montgomery, Alabama
  - Peoria, Arizona
  - Upland, California
  - Colorado Springs, Colorado
  - Brooksville, Florida
  - Inverness, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Savannah, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Overland Park, Kansas
  - Louisville, Kentucky
  - Portland, Maine
  - Rockville, Maryland
  - Billings, Montana
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Eugene, Oregon
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wexford, Pennsylvania
  - Hilton Head Island, South Carolina
  - Midvale, Utah
  - Norfolk, Virginia
  - Richmond, Virginia